CLINICAL TRIAL: NCT05417009
Title: Vagal Autonomic Neuromodulation by Transcutaneous Nerve Stimulation in Acute Ischaemic Stroke Requiring Mechanical Thrombectomy.
Brief Title: Autonomic Neuromodulation by Transcutaneous Nerve Stimulation in Acute Ischaemic Stroke.
Acronym: VANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 314067
Record Dates: First submitted 2022-06-08; First posted 2022-06-14 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke; Thrombotic Stroke; Autonomic Dysfunction; Autonomic Imbalance
MeSH Terms: conditions — Ischemic Stroke; Thrombotic Stroke; Primary Dysautonomias

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham settings for neuromodulation device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation (Active Comparator): Electrodes attached bliaterally to tragus nerve region of outer ear, with appropriate device settings to deliver current.
  Interventions: Device: trans-cutaneous auricular sensory stimulation
- Electrode attachment only. (Sham Comparator): Electrodes attached bliaterally to tragus nerve region of outer ear, with device switched off [blinded to operator].
  Interventions: Device: trans-cutaneous auricular sensory stimulation

INTERVENTIONS:
Device: trans-cutaneous auricular sensory stimulation — Transcutaneous auricular sensory stimulation

SUMMARY:
Autonomic modulation by transcutaneous vagal nerve stimulation in acute ischaemic stroke requiring mechanical thrombectomy: a phase IIa, sham controlled randomised trial.

DETAILED DESCRIPTION:
Loss of autonomic variability is strongly associated with adverse outcomes after ischaemic stroke. Removing blood clots from the brain by mechanical thrombectomy has revolutionised the management of stroke, but more than 50% of patients do not regain functional independence.(PMID:26898852) Blood pressure (BP) control is important, since low and high BP (BP variability) are strongly associated with poor patient outcomes after thrombectomy. (PMIDs:32961389;31964286) Autonomic dysfunction causes labile blood pressure. Intact autonomic function is required to control blood pressure and potentially improve recovery after stroke. Impairment of baroreflex autonomic function, due to reduced vagal activity is associated with extreme BP variability, leading to further brain injury and cardiovascular complications.(PMID:30371208) Reduced baroreflex control is related to poor patient outcomes after stroke, independent of absolute blood pressure.(PMID:19834010) Reversing baroreflex and vagal dysfunction is, therefore, widely held to have the potential to improve cardiovascular control and patient outcome in this context.(PMID:19834010)

Non-invasive peripheral neuromodulation restores autonomic control. Vagal nerve stimulation improves autonomic control and reverses baroreflex dysfunction (PMIDs:28949064) but this has previously required surgically implanted devices which are expensive and impractical in the context of acute stroke. Afferent Electronic have achieved the same effect as these implantable devices by non-invasive transcutaneous autonomic neuromodulation (TAN). We have used this simple, safe, hand-held, low-cost device to increase vagal activity and baroreflex sensitivity through non-invasive, painless stimulation of nerves located in the outer ear to control blood pressure.

Baroreflex sensitivity can be increased at the bedside by TAN for 30 minutes following acute trauma. If this can be replicated in thrombectomy patients, it will aid recovery and rehabilitation through five complementary mechanisms where it has been clinically demonstrated that increasing vagal nerve activity:

1. Restore baroreflex sensitivity;
2. Increase blood flow to ischaemic brain tissue through vagal activation.(PMID:27357059)
3. Dampen cerebral/systemic inflammation.(PMID:26723020);
4. Reduce atrial fibrillation and myocardial injury,(PMIDs:5744003,22739118) which are common after stroke, and independently predict cognitive decline and cardiovascular mortality
5. Allows immediate commencement of vagal nerve stimulation, which has recently been shown to enhance upper-limb rehabilitation.(PMID:33894832) Our proof-of-concept data shows daily TAN reduces BP and BP variability lasting several months even in drug-resistant hypertensive patients. In this proof-of-concept randomised sham-controlled trial, we will examine whether early TAN on presentation for mechanical thrombectomy improves autonomic function in patients with acute ischaemic stroke by reducing blood pressure lability.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing mechanical thrombectomy for acute ischaemic stroke requiring general or sedation.
* Established hypertensive and/or hypertensive on admission for mechanical thrombectomy [systolic BP >140mmHg; diastolic BP >80mmHg]

Exclusion Criteria:

* Current participation in a clinical trial of a treatment with a similar biological mechanism.
* Previous enrolment into VANS trial.
* Anatomical or other contraindication to trans-cutaneous auricular sensory stimulation
* Pregnancy.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gareth L Ackland, PhD FRCA, Principal Investigator — William Harvey Research Institute, Queen Mary University of London
Locations (1):
- William Harvey Research Institute, Barts and The London School of Medicine and Dentistry, Queen Mary University of London, John Vane Science Centre, Charterhouse Square, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Researchers who provide a methodologically sound proposal approved by an independent review committee intermediary using deidentified data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: No end date.
Access Criteria: To achieve aims in approved proposal.

REFERENCES:
- [Derived] Ackland GL, Crane D, Ahuja S, Patel A, Martin T, Joseph M, Ottley O, Hameed R, Dias P, Begum S, Schroth J, Hewson R, Del Arroyo AG, Abbott TEF, Bhogal P. Transauricular Vagus Nerve Stimulation in Acute Ischaemic Stroke Requiring Mechanical Thrombectomy: Sham-Controlled, Randomised Device Trial. Transl Stroke Res. 2025 Dec 27;17(1):10. doi: 10.1007/s12975-025-01404-7. PMID 41455014
- [Derived] Ackland GL, Martin T, Joseph M, Dias P, Hameed R, Gutierrez Del Arroyo A, Hewson R, Abbott TEF, Spooner O, Bhogal P. Transauricular nerve stimulation in acute ischaemic stroke requiring mechanical thrombectomy: Protocol for a phase 2A, proof-of-concept, sham-controlled randomised trial. PLoS One. 2023 Dec 22;18(12):e0289719. doi: 10.1371/journal.pone.0289719. eCollection 2023. PMID 38134136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred for urgent mechanical thrombectomy.
Groups:
- Stimulation - n=18: Electrodes attached bliaterally to tragus nerve region of outer ear, with appropriate device settings to deliver current.
  trans-cutaneous auricular sensory stimulation: Transcutaneous auricular sensory stimulation
- Electrode Attachment Only - n=18: Electrodes attached bliaterally to tragus nerve region of outer ear, with device switched off [blinded to operator].
  trans-cutaneous auricular sensory stimulation: Transcutaneous auricular sensory stimulation
Period: Overall Study
Arm/Group | Stimulation - n=18 | Electrode Attachment Only - n=18
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stimulation - n=18: Electrodes attached bilaterally to tragus nerve region of outer ear, with appropriate device settings to deliver current.
  trans-cutaneous auricular sensory stimulation: Transcutaneous auricular sensory stimulation
- Electrode Attachment Only - n=18: Electrodes attached bilaterally to tragus nerve region of outer ear, with device switched off [blinded to operator].
  trans-cutaneous auricular sensory stimulation: Transcutaneous auricular sensory stimulation
- Total: Total of all reporting groups
Arm/Group | Stimulation - n=18 | Electrode Attachment Only - n=18 | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (13) | 69 (15) | 69 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-white | 8 | 3 | 11
  Other | 10 | 15 | 25
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Variability
Description: Coefficient of variation of systolic blood pressure
Time Frame: 0-24h after mechanical thrombectomy
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Stimulation | Electrode Attachment Only.
Number analyzed (Participants) | 18 | 18
coefficient of variation | 0.106 (0.029) | 0.107 (0.027)

2. Secondary Outcome: Systolic Blood Pressure Variability.
Description: Systolic blood pressure standard deviation.
Time Frame: 0-24h after mechanical thrombectomy
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stimulation - n=18 | Electrode Attachment Only - n=18
Number analyzed (Participants) | 18 | 18
mmHg | 14 (5) | 14 (4)

3. Secondary Outcome: Diastolic Blood Pressure Variability
Description: coefficient of variation- diastolic blood pressure
Time Frame: 24h after admission for mechanical thrombectomy
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Stimulation | Electrode Attachment Only.
Number analyzed (Participants) | 18 | 18
coefficient of variation | 0.136 (0.05) | 0.127 (0.04)

ADVERSE EVENTS:
Time Frame: From randomisation until 7 days after thrombectomy
Description: Daily assessment while in hospital
Arm/Group | Stimulation - n=18 | Electrode Attachment Only - n=18
All-Cause Mortality (participants affected / at risk) | 0/18 | 2/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation - n=18 (N=18) | Electrode Attachment Only - n=18 (N=18)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — local electrode irritation
Anaesthetic complication (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — High airway pressure during mechnical ventilation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT05417009/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT05417009/SAP_001.pdf